CLINICAL TRIAL: NCT03137394
Title: Development of a Biopsychosocial Prospective Surveillance Model of Shoulder Pain in Individuals With Spinal Cord Injury
Brief Title: Development of a Model of Shoulder Pain Following Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Margaret A. Finley, Associate Professor, Drexel University
Other Study IDs: SC160041
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; shoulder pain; psychosocial
MeSH Terms: conditions — Spinal Cord Injuries; Shoulder Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Cord Injury: Participants with SCI in the acute, in-patient rehabilitation phase.Data for each participant in the SCI group will be collected at baseline, 6 months, and 1 year post injury;
  Interventions: Other: Observation
- Able-bodied control: Age- and gender-matched able-bodied individuals (matched to SCI group). Control group data will be collected at baseline and at the 1-year follow-up.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Data for each participant in the SCI group will be collected at baseline, 6 months, and 1 year post injury; control group data will be collected at baseline and at the 1-year follow-up.

SUMMARY:
This study will investigate the progression of musculoskeletal (shoulder muscle flexibility, muscle strength, movement coordination, and rotator cuff health) and psychosocial (fear of movement, pain catastrophizing) impairments for the first year following SCI, starting with inpatient rehabilitation, at 6 months, and at 1 year following SCI.

We will use the information obtained from this study information to develop a biopsychosocial prospective surveillance model, a method for early detection, intervention, and moderation of shoulder pain. Specifically, we will identify sources of biopsychosocial shoulder pain to establish effective physical and cognitive-behavioral treatment to prevent loss of function and independence in individuals with SCI who depend on their arms for activities of daily living, transfers, and wheelchair propulsion.

DETAILED DESCRIPTION:
Shoulder pain is a common secondary condition in people with spinal cord injury (SCI) that often results in loss of function and of independence and imposes limitations on self-care, work, and leisure activities, and leads to decreased quality of life. More than 40% of individuals with SCI report shoulder pain at the beginning of inpatient rehabilitation; this number increases to 50% at hospital discharge. The onset of shoulder pain within the first year after injury may lead to lifelong chronic shoulder pain. Although information is known about shoulder pain in patients with long-term SCI, little is known about the beginning of shoulder problems and how they progress early after the injury. In addition to physical problems, psychosocial factors are also associated with chronic pain.

This study will investigate the progression of musculoskeletal (shoulder muscle flexibility, muscle strength, movement coordination, and rotator cuff health) and psychosocial (fear of movement, pain catastrophizing) impairments for the first year following SCI, starting with inpatient rehabilitation, at 6 months, and at 1 year following SCI. Age- and gender-matched controls will be compared at baseline and at 1 year.

Instead of routinely screening patients to identify and treat related factors before shoulder pain and dysfunction become problems, the current practice is to start treatment after shoulder pain occurs. We will use the information obtained from this study information to develop a biopsychosocial prospective surveillance model, a method for early detection, intervention, and moderation of shoulder pain. Specifically, we will identify sources of biopsychosocial shoulder pain to establish effective physical and cognitive-behavioral treatment to prevent loss of function and independence in individuals with SCI who depend on their arms for activities of daily living, transfers, and wheelchair propulsion. Early identification of problem areas may provide a method to refer a patient for treatment or to change ongoing intervention. Development of a biopsychosocial prospective surveillance model will provide a proactive approach to reduce the debilitating consequences of activity limitations and participation restrictions in individuals with SCI, reducing the burden currently experienced by military service members, veterans, and their families and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible for participation if they are >18 years of age and included in the SCI group if they demonstrate a complete or incomplete SCI of American Spinal Injury Association grade A, B, C or D45; attend inpatient rehabilitation following SCI; use a manual wheelchair for at least 50% mobility; and are medically stable.
* The control group will able-bodied (non-SCI) and be age and sex matched to the SCI group

Exclusion Criteria:

* Individuals will be excluded from participating in either group if they present with upper extremity radicular symptoms; preexisting neurological conditions; and complications from other health conditions that could influence upper extremity function.
* Control group: Individuals will be excluded from participating in any group if they present with preexisting neurological conditions; and complications from other health conditions that could influence upper extremity function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 68 individuals across both sites will be enrolled [34 at each the Drexel site and the University of Maryland Rehabilitation & Orthopaedic Institute (UM Rehab)].
  Participants with SCI will be recruited through the Magee Rehabilitation Hospital network (see letter of support). Individuals without SCI will be recruited from the local community. A member of the research team will serve will identify, screen, and obtain consent from interested, eligible individuals in the group with acute SCI. Individuals for the control group will be recruited with flyers and through personal contact with Magee Rehabilitation Hospital, UMRehab, and the community at large.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal Pain Survey (MPS)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  Change in musculoskeletal pain will be assessed with the self-report Musculoskeletal Pain Survey.[20] This questionnaire asks the person to rate the presence, seriousness, and frequency of pain in the joints or muscles of the upper extremities. A composite pain score is calculated for bilateral upper extremities, ranging from 0 to 90. The shoulder pain score will also be analyzed separately (score 0 to 30). This scale has been used to identify musculoskeletal pain in individuals with SCI.[20-22]
Pectoralis Minor Muscle Length Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  Manual palpation will identify the fourth rib and the coracoid process.[47] Pectoralis minor length will be measured as the distance between the fourth rib and coracoid process under two testing conditions: resting posture and passive lengthening.[48] Pectoralis minor muscle length will be measured as the distance between the two landmarks (cm) with the Palpation Meter (PALM, St. Paul, MN).[47] We have established excellent measurement properties for our procedure of measuring pectoralis minor muscle length under resting and passive lengthening conditions (ICC2,2=0.86-0.94, MDC95 =1.77cm).[49]
Shoulder Girdle Tissue Integrity Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  Musculoskeletal ultrasound with a multifrequency, broadband, 50-mm linear array transducer will be used to obtain images of the subscapularis supraspinatus infraspinatus and biceps tendons, acromiohumeral distance, and supraspinatus muscle fatty infiltrate.5[0] Accuracy of musculoskeletal ultrasound for detection of rotator cuff tears is reported to be 88.9% (95% confidence interval =74.1 to 96.21).[51] Dr. Trojian has extensive training in the use of diagnostic ultrasound of the shoulder complex and will perform the ultrasound examinations. One assessor, masked to participant group and age, will provide the clinical interpretation of the finding and identify changes over time.
Tampa Scale of Kinesiophobia Scale (TSK-11)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  The TSK-11 is used to assess fear of movement (kinesiophobia).41,42 The validated 11-item version (TSK-11)[52] gives a score range of 11 to 44, with higher scores indicating higher fear of movement and reinjury. The TSK -11 comprises opinion-based items that evaluate the participants' general status on a scale of 1 to 4 (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). TSK-11 offers excellent reliability (ICC=0.81, SEM=2.54).5[2]
Fear of Pain Questionnaire (FPQ)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  The FPQ43 is a 30-item measure of fear of painful stimuli. The FPQ includes three subscale scores for minor pain, severe pain, and medical pain. For each painful situation described on the FPQ, participants rate how "fearful" they are on a scale from 1 (not at all) to 5 (extreme). Previous research reported adequate internal consistency (α range, 0.86-0.87) on the FPQ scales.[53]
Pain Catastrophizing Scale (PCS)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  The PCS consists of 13 items rated on a 5-point scale (0=not all to 4=all the time).[27] Participants are instructed to rate the degree to which specified thoughts and feelings occur when experiencing pain. Three dimensions of pain catastrophizing are assessed: rumination, magnification, and helplessness. Only the total score was used in the current study. The PCS is validated for clinical and nonclinical populations.[27,36,53,54]
Subjective Quality of Life Questionnaire (SQoL)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  This questionnaire is a global measure of subjective perception of QoL.[55] The scale is a Likert-type scale measuring satisfaction with life as a whole: Participants are asked to take everything in their life into account and rate it on an ordinal scale from 1 (life is very distressing; it's hard to imagine how it could get much worse) to 7 (life is great; it's hard to imagine how it could get much better).[56] Test-retest reliability is high (91% agreement),[55] and this questionnaire is validated with the SCI population.[55,57,58] Dr. Mulroy holds expertise and experience in using psychosocial measures in individuals with SCI and will oversee the analysis and interpretation of these primary and secondary measures.

SECONDARY OUTCOMES:
Muscle Strength-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  We will collect measures of shoulder girdle muscle abduction, adduction, internal rotation, and external rotation strength. Standard manual muscle testing positions of Kendall et al.[59] will be used when possible; a modification of the position will be used in an effort to perform all tests with participants seated in their wheelchairs. A handheld dynamometer will be used to record the peak muscle force over three trials; the highest value will be used for analysis. Dynamometry is a reliable method for assessing strength (ICC=0.97).60 We will determine muscle strength ratios for abduction/adduction, internal/external rotation, and protraction/retraction.[14]
Chronic Pain Coping Inventory-42 (CPCI-42)-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  The CPCI, a 42-item abbreviated version of the original 65-item CPC [,6]1 asks individuals to self-report the frequency of use of particular behavioral and cognitive strategies to cope with pain; it has good psychometric properties.6[2] Specifically, the CPCI-42 lists coping strategies and asks participants "During the past week, how many days did you use each of the following at least once in the day to cope with your pain?" CPCI scales demonstrate adequate to excellent test-retest stability (0.65-0.90).

OTHER OUTCOMES:
Upper Extremity Kinematic/ Intersegmental Coordination-Change over time | SCI Group: baseline, 6-months, one-year; Control Group: baseline, one-year
  Three-dimensional kinematic data of the trunk, scapula, and humerus will be collected (100 Hz) during a functional overhead reaching task with the Motion Monitor electromagnetic transmitter system (Innovative Sports Training, Inc., Chicago, IL).[63] Sensor placement and global and local coordinate system definitions will be based on the International Society of Biomechanics recommendations for shoulder kinematics. [64] Coupling angles and phase-angle analysis will determine intersegmental coordination of the scapula and humerus throughout the range of humerothoracic elevation. Drs. Finley and Ebaugh have extensive experience in biomechanical analysis of 3-dimensional shoulder girdle kinematics and will collect and interpret the kinematic data.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Finley, PT,PhD, Principal Investigator — Drexel University
Locations (2):
- United States (2):
  - University of Maryland Rehabilitation and Orthopedic Institute, Gwynn Oak, Maryland
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Results will be presented at annual meetings, as described below as well as anticipated numerous manuscripts, regardless of the results. The outcomes will be of interest to the public, researchers, policy makes, and funding sources. Final Research Data (de-identified and unidentifiable) defined as recorded factual material commonly accepted in the scientific community as necessary to document and support research findings will be available upon request of such agencies as the DOD, the Food and Drug Administration (FDA), Medicare/Medicaid, or others who hold interest or cause to review the raw data. No protected health information (PHI) will be collected for this study.

REFERENCES:
- [Background] Finley M, Euiler E, Baehr L, Gracely E, Brownsberger M, Schmidt-Read M, Frye SK, Kallins M, Summers A, York H, Geigle PR. Relationship of psychosocial factors and musculoskeletal pain among individuals with newly acquired spinal cord injury. Spinal Cord Ser Cases. 2021 Jul 19;7(1):61. doi: 10.1038/s41394-021-00415-4. PMID 34282128
- [Background] Finley M, Euiler E, Trojian T, Gracely E, Schmidt-Read M, Frye SK, Kallins M, Summers A, York H, Geigle PR. Shoulder impairment and pain of individuals with newly acquired spinal cord injury compared to uninjured peers. Spinal Cord Ser Cases. 2020 Aug 4;6(1):68. doi: 10.1038/s41394-020-0318-1. PMID 32753624
- [Background] Finley MA, Euiler E, Hiremath SV, Sarver J. Movement Coordination During Humeral Elevation in Individuals With Newly Acquired Spinal Cord Injury. J Appl Biomech. 2020 Aug 14;36(5):345-350. doi: 10.1123/jab.2019-0387. Print 2020 Oct 1. PMID 32796138